CLINICAL TRIAL: NCT06138340
Title: The Alterations of Brain Network Connectivity Under Sedation and Anesthesia in Patients With Supratentorial Glioma
Brief Title: The Effects of Anesthetics on Brain Network Connectivity in Patients With Supratentorial Glioma
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Deputy chief of Department of Anesthesiology, Beijing Tiantan Hospital
Other Study IDs: 20230808
Record Dates: First submitted 2023-09-11; First posted 2023-11-18 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Brain Network Connectivity; Postoperative Delirium; Dexmedetomidine; Propofol
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Propofol; remimazolam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dex group: Participants will be sedated and maintained by dexmedetomidine.
  Interventions: Drug: Dexmedetomidine
- Propofol group: Participants will be sedated and maintained by propofol.
  Interventions: Drug: Propofol
- Remimazolam group: Participants will be sedated and maintained by remimazolam.
  Interventions: Drug: Remimazolam Injection

INTERVENTIONS:
Drug: Dexmedetomidine — Participants will be sedated and maintained by dexmedetomidine during the surgery.
  Groups: Dex group
Drug: Propofol — Participants will be sedated and maintained by propofol during the surgery.
  Groups: Propofol group
Drug: Remimazolam Injection — Participants will be sedated and maintained by remimazolam during the surgery.
  Groups: Remimazolam group

SUMMARY:
Perioperative anesthesia can affect postoperative cognitive function. In our previous study, intraoperative dexmedetomidine (Dex) infusion reduced the incidence of delirium within the first 5 days after brain tumor. However, the mechanism is still unclear. With the development of neuroimaging, multimodal neuroimaging technology provide a new method to explore the underlying mechanism. Therefore, the purpose of this study is to analyze the alterations of brain network under sedation and anesthesia by different anesthetics in patients with supratentorial glioma and their association with cognition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as unilateral supratentorial glioma by MRI
* Selective operation
* Age over 18 years old
* ASA I-II
* Right handedness

Exclusion Criteria:

* History of cerebrovascular disease, brain trauma, chemotherapy and radiotherapy, or psychotropic drugs
* History of intracranial surgery
* Drug and/or alcohol abuse
* History of dementia or mental illness
* Pregnant or lactating women
* Contraindications for MRI
* Severe bradycardia (heart rate less than 40 beats per minute), sick sinus syndrome or second-to-third degree atrioventricular block
* Severe hepatic or renal dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be selected from patients who schedule to receive elective surgery in Beijing Tiantan Hospital.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The alterations of brain network connectivity. | Before sedation, 30 minutes after sedation，and 30 minutes after surgery.
  fMRI and DTI will be used to detect brain network connectivity.

SECONDARY OUTCOMES:
Postoperative delirium. | Day 1-5 after surgery.
  The incidence and severity of postoperative delirium and its association with changes of brain network connectivity.
Electroencephalogram changes | From patients admission to operation room until 10 minutes after surgery
  Electroencephalogram will be used to record the brain activity.
rScO2 changes. | From patients admission to operation room until 10 minutes after surgery
  Regional cerebral oxygen saturation (rScO2) will be monitored with near-infrared spectroscopy (NIRS).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality, China